CLINICAL TRIAL: NCT05205408
Title: A Single-Arm, Open-Label, Dose Escalation Study to Evaluate Safety and Efficacy of Intratumoral Injection of Oncolytic Virus Injection (RT-01) in Patients With Advanced Solid Tumors
Brief Title: A Study of Intratumoral Administration of Oncolytic Virus Injection (RT-01) in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Wang Zishu, Director of the Department of Medical Oncology, The First Affiliated Hospital of Bengbu Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LWY21076CBY1
Record Dates: First submitted 2022-01-19; First posted 2022-01-25 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumor
Keywords: RT-01; Oncolytic Virus; immunotherapy; Intratumoral injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic Virus Injection(RT-01) (Experimental): Intratumoral administration of RT-01 as single agent for patients with advanced solid tumors. Dose cohorts: 1×10^8 TCID50/mL and 7×10^8 TCID50/ mL
  Interventions: Biological: Oncolytic Virus Injection(RT-01)

INTERVENTIONS:
Biological: Oncolytic Virus Injection(RT-01) — Administered by intratumoral injection as single agent.

SUMMARY:
This is a single-arm, open-label, dose escalation, clinical pharmacology study to evaluate safety and efficacy of oncolytic virus injection(RT-01) When Administered Via Intratumoral Injection in patients with advanced solid tumors.

The primary purpose of this study is to evaluate the safety and tolerability, the secondary purpose is to evaluate the antitumor activity, immunoreactivity, immunogenicity, pharmacokinetics and virus shedding of RT-01.

DETAILED DESCRIPTION:
This is an investigator initiated , single-arm, open-label, dose escalation clinical pharmacology study of RT-01 as a single agent given via Intratumoral injection in patients with advanced solid tumors.

The study is a single agent dose escalation which will use an accelerated and "3+3" design to evaluate escalating doses of RT-01. Total enrollment will depend on the toxicities and/or activity observed, with approximately 6-12 evaluable participants enrolled. A Dose-Limiting Toxicity (DLT) observation period of 4 weeks was established before the entry of the first patient at the next dose level.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years;
* Subjects must have histologically or cytologically confirmed diagnosis of advanced solid tumor(s) who have failed in standard therapy (disease progression or intolerance) and no effective treatment, or have no standard therapy, or have failed to obtain standard treatment due to objective conditions;
* Subjects have At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
* ECOG score of 0 ~ 2;
* Adequate bone marrow, hepatic and renal and coagulation function;
* Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
* Voluntarily participated in this study, signed the informed.

Exclusion Criteria:

* Subjects with known brain metastasis and/or clinically history tumor brain of metastasis;
* Subjects who have received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc within 2 weeks before RT-01 administration;
* Subjects who have participate in another interventional study within 4 weeks before RT-01 administration;
* Subjects who have had major surgery within 4 weeks before RT-01 administration;
* Patients in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days before RT-01 administration, but currently or previously treated with any of the following steroid regimens, were included: Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption; Prophylactic short-term use of corticosteroids;
* Subjects who have participate in another oncolytic virus study within 8 weeks before RT-01 administration;
* Subjects received live vaccines within 7 days before RT-01 administration;
* Subjects received Antiviral drugs within 2 weeks, long-acting interferon within 4 weeks before RT-01 administration;
* Subjects with adverse reactions caused by previous anti-tumor treatment not recovered to (CTCAE 5.0) grade 1 (except alopecia);
* Subjects who have uncontrolled active infection;
* Subjects with known positive history of human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS);
* Subjects who have active hepatitis;
* Subjects who have serious cardiovascular system disorders history;
* Subjects with active autoimmune diseases or history of autoimmune diseases that may relapse;
* Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator;
* Subjects in other conditions that are considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Up to 28 days
  Dose-limiting toxicity is defined as an adverse event that is considered to be drug-related and meets one of the Protocol definitions

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.
To evaluate the antitumor activity. | Up to 2 years
  Assessed per RECIST and iRECIST
The changes of the immunoreactivity during treatment | Up to 28 days
  Peripheral blood T lymphocyte subtype
To evaluate the immunogenicity of RT-01 | Up to 28 days
  Antiviral antibody
To evaluate the viral shedding of RT-01 | Up to 24 Weeks
  Viral RNA
The Pharmacokinetics characteristics of RT-01 | Up to 24 Weeks
  The Cmax of Viral RNA
The Pharmacokinetics characteristics of RT-01 | Up to 24 Weeks
  The Tmax of Viral RNA

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No